CLINICAL TRIAL: NCT03281382
Title: PHASE 1 TRIAL OF ONCOLYTIC ADENOVIRUS-MEDIATED CYTOTOXIC AND IL-12 GENE THERAPY IN COMBINATION WITH CHEMOTHERAPY FOR THE TREATMENT OF METASTATIC PANCREATIC CANCER
Brief Title: Phase 1 Trial of Interleukin 12 Gene Therapy for Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David Kwon, MD, Medical Director, Center for Cancer Surgery, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11260
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Investigational Arm (Experimental): Patients will receive a single intratumoral injection of the oncolytic Ad5-yCD/mutTKSR39rep-hIL12 adenovirus at one of three dose levels. Two days later, subjects will be administered (orally) 7 days of 5-fluorocytosine (5-FC) prodrug therapy. Fourteen days after completion of the 5-FC prodrug therapy course, subjects will be administered chemotherapy at the discretion of the treating physician. On an optional basis, subjects will be administered [18F]-FHBG, a HSV-1 TK substrate, and will undergo PET imaging to quantify the intensity, persistence, and biodistribution of HSV-1 TK gene expression in the pancreas.
  Interventions: Biological: Ad5-yCD/mutTKSR39rep-hIL12

INTERVENTIONS:
Biological: Ad5-yCD/mutTKSR39rep-hIL12 — Oncolytic adenovirus expressing two suicide genes and human IL-12

SUMMARY:
This phase 1 trial will investigate the toxicity of combining interleukin 12 gene therapy with standard chemotherapy in metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This protocol proposes a phase 1 trial combining oncolytic adenovirus-mediated cytotoxic and IL-12 gene therapy with chemotherapy in metastatic pancreatic cancer. Nine subjects (3 cohorts, 3 subjects/cohort) with metastatic pancreatic cancer will receive a single intratumoral injection of the oncolytic Ad5-yCD/mutTKSR39rep-hIL12 adenovirus at one of three dose levels (cohort 1- 1 x 1011 vp, cohort 2- 3 x 1011 vp, cohort 3- 1 x 1012 vp). Depending on the location of the target lesion, the adenovirus will be injected either through the stomach or duodenal wall using endoscopic ultrasound (EUS) guidance. Two days later, subjects will be administered (orally) 7 days of 5-fluorocytosine (5-FC) prodrug therapy. Fourteen days after completion of the 5-FC prodrug therapy course, subjects will be administered chemotherapy at the discretion of the treating physician. On an optional basis, subjects will be administered [18F]-FHBG, a HSV-1 TK substrate, and will undergo PET imaging to quantify the intensity, persistence, and biodistribution of HSV-1 TK gene expression in the pancreas.

The primary endpoint is toxicity at day 21. A secondary endpoint is rates of ≥ grade 3 CTCAE adverse events. Exploratory endpoints include 1) intensity, persistence, and biodistribution of HSV-1 TK gene expression, and 2) association of immunological measurements (i.e., cytokine levels, NK cytolytic activity) with toxicity and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven (biopsy or cytology) metastatic pancreatic adenocarcinoma.
* Age ≥ 18 years.
* No prior treatment (surgery, chemotherapy, radiotherapy, or biological therapy) for the study cancer.
* Zubrod performance score of 0 - 2 within 30 days of registration.
* Subjects must have adequate baseline organ function, as assessed by the following laboratory values, within 30 days before initiating the study therapy:

  * Adequate renal function with serum creatinine ≤ 1.8 mg/dL or creatinine clearance ≥ 50 mL/min/m2.
  * Absolute neutrophil count > 1,000/μL.
  * Hemoglobin > 8.0 g/dL.
  * Platelet count > 100,000/μL.
  * Bilirubin < 2.0 mg/dL.
  * SGOT and SGPT < 3.0 times upper limit of normal (ULN). Subjects with liver metastases may have SGOT/SGPT < 5.0 times ULN.
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout and for 60 days beyond the treatment phase of the study.
* Subjects on oral warfarin anticoagulation therapy may be included in this study, but must have close monitoring of their coagulation parameters as altered parameters and/or bleeding have been reported in patients taking Xeloda® and such agents concomitantly. Subjects on other forms of anti-coagulation therapies may need close clinical monitoring for signs or symptoms of bleeding.
* The subject must possess the ability to give informed consent and express a willingness to meet all of the expected requirements of the protocol for the duration of the study.

Exclusion Criteria:

* Pregnant and lactating women.
* Clinical or laboratory evidence of pancreatitis, based on discretion of treating physician.
* Serious non-malignant disease (e.g., congestive heart failure or uncontrolled infections), which, in the opinion of the investigator would compromise study objectives.
* Major surgery planned within 3 months of registration other than diagnostic procedures such as laparoscopy or endoscopic ultrasound and stenting or PEG/PEJ placement.
* Islet cell tumor, benign cyst, peri-ampullary carcinoma or any non-adenocarcinomas.
* Acute infection. Acute infection is defined by any viral, bacterial, or fungal infection that has required specific therapy within 72 hours of initiation of the study therapy (defined as day 1).
* Previous history of liver disease including hepatitis.
* Positive serologic test for Hepatitis B or C at baseline.
* Immunosuppressive therapy including systemic corticosteroids. Use of inhaled and topical corticosteroids is permitted.
* Impaired immunity or susceptibility to serious viral infections.
* Allergy to any product used on the protocol.
* Serious medical or psychiatric illness or concomitant medication, which, in the judgment of the investigator, might interfere with the subject's ability to respond to or tolerate the treatment or complete the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Toxicity of the gene therapy | 21 days
  grade 1 - 5 CTCAE adverse events

SECONDARY OUTCOMES:
>= grade 3 adverse events | 21 days
  grade 3 - 5 CTCAE adverse events
PET imaging | 14 days
  HSV-1 TK gene expression via [18F]-FHBG administration and PET imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No